CLINICAL TRIAL: NCT00110630
Title: Smoking Treatment of Prisoners: Project "STOP"
Brief Title: Smoking Treatment of Prisoners
Acronym: STOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Karen Cropsey, Univeristy of Alabama at Birmingham
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-15774-2; K23-15774-2
Record Dates: First submitted 2005-05-11; First posted 2005-05-11 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-09

CONDITIONS: Tobacco Use Cessation; Tobacco Use Disorder
Keywords: nicotine dependence
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: 10-week smoking cessation group therapy combined with NicoDerm CQ

SUMMARY:
The purpose of this study is to determine the efficacy of a 10-week smoking cessation therapy combined with NicoDerm CQ for smoking cessation among female prisoners.

DETAILED DESCRIPTION:
This is a randomized controlled trial utilizing a wait-list control group to examine 10-week group therapy and nicotine replacement compared to wait-list for smoking cessation among female prisoners.

ELIGIBILITY:
Inclusion Criteria:

* 1) current smoker and (2) seeking group treatment to quit smoking.

Exclusion Criteria:

* (1) non-english speaking, (2) housed in segregation, (3) presence of active, severe mental illness as defined by active psychosis, manic episode, or imminently suicidal/homicidal, (4) mental retardation such that they cannot provide informed consent, and (5) due to be released or transferred to another facility within the next year.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2005-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
smoking cessation

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cropsey, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States